CLINICAL TRIAL: NCT06061601
Title: Use of a Lower Limb Exoskeleton in Locomotor Rehabilitation of Stroke Patients: Feasibility, Safety and a Pilot Clinical Study
Brief Title: ACTive Exoskeleton for Unilaterally-Assisted Locomotion (ACTUAL)
Acronym: ACTUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: ESOFDG-IIT 2.0
Record Dates: First submitted 2023-07-04; First posted 2023-09-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Stroke Sequelae; Gait, Hemiplegic
Keywords: User centered design; Stroke; Gait rehabilitation; Hemiparesis; Exoskeleton
MeSH Terms: conditions — Gait Disorders, Neurologic; Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: A pilot intervention feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exoskeleton Stroke group (Experimental): This group will receive gait rehabilitation with the exoskeleton for 20 sessions in clinic.
  Interventions: Device: Exoskeleton stroke group
- Healthy control group (No Intervention): The quantitative data, including EMG and 3D kinematics, from 10 healthy controls walking with the exoskeleton will serve as comparative data for the experimental group.

INTERVENTIONS:
Device: Exoskeleton stroke group — The exoskeleton stroke group will receive gait rehabilitation with the TWIN-Acta exoskeleton
  Other Names: TWIN-Acta exoskeleton
  Arms: Exoskeleton Stroke group

SUMMARY:
Walking difficulties are common symptoms after stroke, significantly reducing quality of life. Walking recovery is therefore one of the main priorities of rehabilitation. Wearable powered exoskeletons have been developed to provide lower limb assistance and enable training for persons with gait impairments by using typical physiological movement patterns. Exoskeleton were originally designed for individuals without any walking capacities, such as subjects with a complete spinal cord injury. Recent systematic reviews suggested that lower limb exoskeletons could be valid tools to restore independent walking in subjects with residual motor function, such as persons post-stroke.The aim of the study was to identify the end-users needs and to develop a user-centered-based control system for the TWIN lower limb exoskeleton to provide an efficient post-stroke rehabilitation of gait. The investigators thus carried out the development and validation through evaluation sessions performed on healthy clinical experts and persons with stroke to evaluate TWIN-Acta usability, acceptability, and barriers of usage. A phase two includes a pilot study of efficacy of using the TWINActa for gait rehabilitation for persons with stroke.

DETAILED DESCRIPTION:
The aim of the study was to identify the end-users needs and to develop a user-centered-based control system for the TWIN lower limb exoskeleton to provide post-stroke rehabilitation. The investigators thus carry out the development and validation of TWIN-Acta: a novel control suite for TWIN, specifically designed for gait rehabilitation of persons post stroke through use of typical physiological movement patterns.

The study will be carried out in two phases. In the first user-centered developmental phase data on usability, acceptability, and limitations to system usage will be collected from clinical experts and persons with stroke through questionnaires and semi-structured interviews.This developmental phase will follow a user-centered approach: it will be based on focus group sessions with clinical and biomechanical experts to define the design specifications for the new control modality of the exoskeleton; consequently evaluation sessions consisting of physical testing of the TWIN-Acta will be carried out by healthy clinical experts and persons with stroke to evaluate TWIN-Acta usability, acceptability, and barriers of usage.

In the second phase of the study a pilot study including 20 sessions of gait rehabilitation of persons at least three month post stroke will be carried out in clinic with the TWIN exoskeleton including the TWIN-Acta control suite.

Outcomes will be verified at baseline and following the intervention through feasibility measures, patient reported outcomes, clinical measures of gait ability and through EMG and 3D gait analysis. The quantitative values will be compared to data of healthy controls walking in the exoskeleton in one session but not receiving any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

  * Age 30-75 anni;
  * 50 kg ≤ weight ≤90 kg
  * 150 cm ≤ height ≤ 192 cm
  * Thigh length: 355 ÷ 475 mm;
  * Length of tibia: 405 ÷ 485 mm;
  * Width pelvis: 690 ÷ 990 mm;
  * Shoe number: 36 ÷ 45
* Subjects with stroke

  * Age 30-75 anni;
  * 50 kg ≤ Weight ≤90 kg
  * 150 cm ≤ Height ≤ 192 cm
  * Thigh length: 355 ÷ 475 mm;
  * Length of tibia: 405 ÷ 485 mm;
  * Pelvic width: 690 ÷ 990 mm;
  * Shoe number: 36 ÷ 45;
  * Stroke diagnosis at least 3 months and within 24 months;
  * First unilateral haemorrhagic or ischemic stroke classified as complete or partial infarction of the anterior circulation and infarction of the lacunar circulation (Oxford Stroke Classification: TACS -Total Anterior Circulation Stroke, PACS - Partial Anterior Circulation Stroke, LACS -Lacunar Stroke). These criteria may include hemiplegia, hemianopia, motor and/or sensory deficits, and disturbance/impairment of superior cortical and subcortical function;
  * FAC (Functional Ambulation Category) 1, 2 and 3 (subjects with ambulation dependent on supervisor or continuous or intermittent physical assistance);
  * At least MRC (Medical Research Council) of the triceps surae equal to 1 or greater (required to produce the biofeedback tone or for exoskeleton control).

Exclusion Criteria:

* Healthy subjects

  * Prosthetic implants
  * Musculoskeletal, neurological, cardiovascular and pulmonary disorders that may impair gait;
  * State of pregnancy or breastfeeding.

Exclusion criteria

* Subjects with stroke

  * Mini Mental State Examination < 23/30;
  * Clinical records of visuospatial and ideomotor apraxia, behavioral disorders (e.g. depression, aggression), neglect, major visual impairment and severe osteoporosis;
  * Non stabilized fractures;
  * Cranial injury;
  * Other diseases attributable to cardio-respiratory problemsi;
  * State of pregnancy or breastfeeding;
  * Previous or concurrent neoplastic malignancy;
  * Chronic inflammatory diseases with joint involvement of the lower limbs;
  * Serious spasticity (Ashworth>3);
  * Pelvic fractures and unstable column;
  * Significant limitations of passive ROM of hips and knees;
  * Problems with skin integrity at the interface surfaces with the device or that would prevent sitting.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in meters walked during the Two minute walking test | Baseline (T0) and after 4 weeks (T1) and after 3 months (T2)
  The subjects were instructed to walk at their usual speed for 2 minutes while the distance they covered in 2 minutes was recorded in meters.

SECONDARY OUTCOMES:
Change in score on the Ashworth scale | Baseline (T0) and after 4 weeks (T1)
  The Ashworth Scale measures muscle resistance during passive limb movement. Minimum and maximum values 0 No increase in muscle tone.
  1. Slight increase in muscle tone, manifested by a minimal stop or resistance at the end of passive movement 1+ Slight increase in muscle tone, manifested by a stop followed by minimal resistance
  2. More marked increase in muscle tone
  3. Considerable increase in muscle tone
  4. Rigid limb in flexion or extension Interpretation of Scores
  0 No increase in muscle tone The resistance perceived towards the end of the movement
  1+ Slight resistance perceived in the first half of the movement 2 Stronger resistance throughout the entire range of motion, but passive movement remains relatively easy.
  3 Substantial resistance, with difficulty in moving the limb passively. 4 The limb is rigid and cannot be moved passively, indicating severe spasticity.
Change in score on the Muscle Manual Test (MMT) | Baseline (T0) and after 4 weeks (T1)
  MMT, is a procedure used to assess a patient's muscle strength on a scale ranging from 0 to 5.
  Minimum and maximum values 0 No visible or palpable contraction.
  1. Visible or palpable muscle contraction
  2. Movement possible but not against gravity
  3. Movement possible against gravity
  4. Movement possible against a certain resistance
  5. Complete muscle strength, normal Interpretation of Scores
  0 Indicates complete paralysis of the evaluated muscle
  1. Indicates minimal muscle activity without joint movement
  2. Indicates significant weakness
  3. Indicates that the patient can move the limb against gravity, but without additional resistance.
  4. Indicates good but not complete muscle strength; the patient can resist a certain resistance, but not maximum.
  5. Indicates complete muscle strength, where the patient can perform movement against full resistance without problems.
Change in time (sec) taken to Timed up and Go | Baseline (T0) and after 4 weeks (T1)
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
Change time (sec) taken to complete the Five time sit to stand (5xSTS) | Baseline (T0) and after 4 weeks (T1) and after 3 months (T2)
  The 5xSTS measures the amount of time it takes for a patient to sit and stand five times in succession with arms folded across their chest.
Change in score on the Stroke impact Scale (SIS) questionnaire | Baseline (T0) and after 4 weeks (T1) and after 3 months (T2)
  The Stroke Impact Scale (SIS) is a tool used to assess the outcome and impact of a stroke on different areas of a patient's life Minimum and maximum values Strength 0-100 Memory and thinking 0-100 Emotions 0-100 Communication 0-100 Activities of daily life 0-100 Mobility 0-100 Social participation 0-100 Interpretation of Scores 0 indicates the worst possible condition or complete disability. 100 represents the best possible state or absence of disability. The higher the score in a given domain, the better the function or well-being perceived by the patient in that area. For example, a high score in the "Mobility" domain indicates that the patient has a good ability to move independently, while a low score may indicate significant difficulties.
Change in time (sec) taken to complete the 10 meter walking test (10mwt) | Baseline (T0) and after 4 weeks (T1) and after 3 months (T2)
  The 10 meters walking test (10MWT) is a test in which the participant is timed while walking 10m at their comfortable speed.
Changes in movement parameters extracted from the kinematics of the body. | Baseline (T0) and after 4 weeks (T1)
  Kinematics of the lower limb will be recorded using a 9 camera optoelectronic system during 3D motor acts.
  The system will measure the 3D coordinates of spherical markers attached to body landmarks to compute hip, knee and ankle angles.
  Data processing will provide measures of deviations from physiological movement.
Correlation between brain activity parameters and motor activity parameters | Baseline (T0) and after 4 weeks (T1)
  Brain activity data acquired with electroencephalogram (EEG) correlated with data from electromyographic systems.
  Data processing will provide measures of deviations from physiological movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Carlo Gnocchi IRCCS, Milan, Italy